CLINICAL TRIAL: NCT01828268
Title: Metabolic Fingerprintings and Metabolic Dynamics After HIV Infection:Impact of Metabolic Changes and Anti-Retroviral Therapy, Life Style and Clinical Conditions
Brief Title: Metabolomics Fingerprinting and Metabolic Dynamics After HIV Infection
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sichuan Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: META-HA-001-2013
Record Dates: First submitted 2013-04-05; First posted 2013-04-10 (Estimated); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: HIV
Keywords: HIV; Metabolomics Fingerprinting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma from peripheral blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- HIV infectors: 100 confirmed HIV-1 infected patients who meet inclusion criteria.

SUMMARY:
The purpose of this plot study is to find out the relationship between metabolic changes and anti-retroviral therapy (ART), life style and clinical conditions of HIV-infected patients using nuclear magnetic resonance (NMR) based systems biology approach and metabolomics methodology.

DETAILED DESCRIPTION:
Since the clinical application of anti-retroviral therapy (ART) in 1997, the life expectancy of HIV infected patients has been prolonged greatly. However,side effects of ART including metabolic abnormalities have become the main factors influencing patients' quality of life. Among which the abnormal lipid metabolism plays an important role. Meanwhile, metabolic conditions differ from patients applying to different combinations of ART drugs,life style and clinical conditions.

Metabolomics can measure the dynamic metabolic responses of the body to stimuli or modifications. Using nuclear magnetic resonance (NMR) as tools can systematically analyse the process of lipid metabolism. Metabolomics fingerprinting can be defined as the complete complement of small molecule (< 1500 Da) metabolites found in a specific cell, body fluid, organ or organism.

Therefore, the study of the impact of metabolic changes and anti-retroviral therapy (ART), life style and clinical conditions is of importance in enhancing the adherence and improving the clinical outcomes of HIV infected patients.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of HIV infection

Exclusion Criteria:

* Pregnancy
* Individual who is participating in other trial(s)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Recruit 100 HIV-infected individuals from community HIV Clinic and/or Transmitted Disease Hospital of Chengdu
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2013-03; Primary Completion 2019-03 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Dyslipidemia | Dyslipidemia events from admission to discharge(Up to 6 months) )

SECONDARY OUTCOMES:
Lipoatrophy | Lipoarophy events from admission to discharge (up to 6 months)

CONTACTS AND LOCATIONS:
Overall Officials: Hua JIANG, PhD, Study Chair — 3Sichuan Academy of Medical Science, Sichuan Provincial People's Hospital, East Branch, Metabonomics and Multidisciplinary Laboratory; Jin PENG, Master, Principal Investigator — 3Sichuan Academy of Medical Science, Sichuan Provincial People's Hospital, East Branch, Metabonomics and Multidisciplinary Laboratory
Locations (1):
- Sichuan Academy of Medical Sciences,Sichuan Provincial Hospital, Metabolomics and Mutidisciplinary Laboratory, Chengdu, Sichuan, China

REFERENCES:
- [Background] Schackman BR, Scott CA, Sax PE, Losina E, Wilkin TJ, McKinnon JE, Swindells S, Weinstein MC, Freedberg KA. Potential risks and benefits of HIV treatment simplification: a simulation model of a proposed clinical trial. Clin Infect Dis. 2007 Oct 15;45(8):1062-70. doi: 10.1086/521933. Epub 2007 Sep 4. PMID 17879926
- [Background] Joly V, Flandre P, Meiffredy V, Leturque N, Harel M, Aboulker JP, Yeni P. Increased risk of lipoatrophy under stavudine in HIV-1-infected patients: results of a substudy from a comparative trial. AIDS. 2002 Dec 6;16(18):2447-54. doi: 10.1097/00002030-200212060-00010. PMID 12461419
- [Background] John M, McKinnon EJ, James IR, Nolan DA, Herrmann SE, Moore CB, White AJ, Mallal SA. Randomized, controlled, 48-week study of switching stavudine and/or protease inhibitors to combivir/abacavir to prevent or reverse lipoatrophy in HIV-infected patients. J Acquir Immune Defic Syndr. 2003 May 1;33(1):29-33. doi: 10.1097/00126334-200305010-00005. PMID 12792352
- [Background] Zhang F, Dou Z, Ma Y, Zhao Y, Liu Z, Bulterys M, Chen RY. Five-year outcomes of the China National Free Antiretroviral Treatment Program. Ann Intern Med. 2009 Aug 18;151(4):241-51, W-52. doi: 10.7326/0003-4819-151-4-200908180-00006. PMID 19687491
- [Background] Zyromski NJ, Mathur A, Gowda GA, Murphy C, Swartz-Basile DA, Wade TE, Pitt HA, Raftery D. Nuclear magnetic resonance spectroscopy-based metabolomics of the fatty pancreas: implicating fat in pancreatic pathology. Pancreatology. 2009;9(4):410-9. doi: 10.1159/000199436. Epub 2009 May 19. PMID 19451751
- [Result] Friis-Moller N, Weber R, Reiss P, Thiebaut R, Kirk O, d'Arminio Monforte A, Pradier C, Morfeldt L, Mateu S, Law M, El-Sadr W, De Wit S, Sabin CA, Phillips AN, Lundgren JD; DAD study group. Cardiovascular disease risk factors in HIV patients--association with antiretroviral therapy. Results from the DAD study. AIDS. 2003 May 23;17(8):1179-93. doi: 10.1097/01.aids.0000060358.78202.c1. PMID 12819520